CLINICAL TRIAL: NCT05787418
Title: A Phase III, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of HH-120 Nasal Spray for Post-exposure Prophylaxis of SARS-CoV-2
Brief Title: HH-120 Nasal Spray for Post-exposure Prevention of SARS-CoV-2
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Huahui Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HH120-NS311
Record Dates: First submitted 2023-03-27; First posted 2023-03-28 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
Keywords: Severe Acute Respiratory Syndrome Coronavirus 2; Coronavirus disease 2019
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HH-120 group (Experimental): HH-120 Nasal Spray
  Interventions: Drug: HH-120 Nasal Spray
- Control group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HH-120 Nasal Spray — HH-120 nasal spray 8 times per day for 7 consecutive days
  Arms: HH-120 group
Drug: Placebo — Placebo 8 times per day for 7 consecutive days
  Arms: Control group

SUMMARY:
This study will assess the efficacy of HH-120 nasal spray in participants for the post-exposure prevention of SARS-CoV-2.

DETAILED DESCRIPTION:
During this study, participants will receive HH-120 nasal spray treatment for 7 consecutive days, the efficacy and safety of HH-120 nasal spray will be assessed throughout the study period mainly based on the incidence of symptomatic SARS-CoV-2 infection and adverse events, respectively.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 85 years old.
* Participants with potential exposure to index patients (with known positive result of qRT-PCR or rapid antigen test [RAT]).
* Participants will be randomized no longer than 48 hours from the onset of the COVID-19 related symptom of the index patients.
* Participants with a negative RAT result within 2 hours prior to randomization.
* Fertile participants must agree to use a highly effective method of contraception.
* Participants being able and willing to provide informed consent prior to any study-specific procedure.

Exclusion Criteria:

* Those with high risk of cardiac events, or severe abnormal functions of liver, kidney, lung, brain and other organs and are deemed as unsuitable to participate in the study (except for those subjects with kidney failure but received regular dialysis, or those with liver dysfunction but stabilized after treatment evaluated by the evaluation of the investigators).
* Those comorbid with asthma.
* Those with a history of SARS-CoV-2 infection within 3 months prior to randomization.
* Those who has received any nasal spray or aerosol inhalation COVID-19 vaccine within 3 months prior to randomization.
* Those who experienced symptom of upper respiratory tract infection within 2 weeks prior to randomization, such as nasal congestion, sore throat, shortness of breath (dyspnea), cough, fatigue, fever, headache, etc.
* Known history of allergy or reaction to any component of the study drug formulation.
* Those who has received other treatment with anti-COVID-19 indication (within 1 month or 5 half-life period prior to randomization, whichever occurs first).
* Participants with nasal disease that is inconvenient or intolerant of nasal spray administration.
* Other reasons considered by the investigator to be unsuitable for the study.

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of symptomatic SARS-CoV-2 infection | Up to 7 days
  Incidence of participants with quantitative Real-Time polymerase chain reaction (qRT-PCR) confirmed SARS-CoV-2 infection and COVID-19 related symptom

SECONDARY OUTCOMES:
The incidence of SARS-CoV-2 infection | Up to 7 days
The changes in SARS-CoV-2 viral nucleic acid load | Up to 7 days
The change of viral load by qRT-PCR | Up to 7 days
Incidence and severity of adverse events | Up to 21 days
The incidence of symptomatic SARS-CoV-2 infection | Up to 3 days
The incidence of symptomatic SARS-CoV-2 infection | Up to 5 days
Time to onset of first COVID-19 related symptom | Up to 7 days
Proportion of participants who progress to moderate/severe/critical type of COVID-19 or death | Up to 21 days
The incidence of symptomatic SARS-CoV-2 infection in different subgroups | Up to 7 days
The incidence and titer of antidrug antibody (ADA) | Up to 21 days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Ditan Hospital, Capital Medical University, Beijing
  - Huashan Hospital of Fudan University, Shanghai